CLINICAL TRIAL: NCT03551041
Title: The Different Neural Representation of Self in Depression Patients and Healthy Individuals.
Brief Title: The Neural Representation of Self in Depression Patients
Status: Completed | Type: Observational
Sponsor: Beijing Normal University (Other)
Collaborators: Peking University (Other); Southwest Medical University (Other)
Responsible Party: Principal Investigator, ma, yina, Professor, Beijing Normal University
Other Study IDs: DepressionSelf_fMRI
Record Dates: First submitted 2018-02-04; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-02

CONDITIONS: Depression Disorder; Healthy
Keywords: depression, self-referential, neural representation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To be aware of oneself as a unique entity in the world occurs early in human development and is the prerequisite of normal social functioning. The disturbance of self representation characterizes a variety of mental disorders such as autism and schizophrenia. Negative self-bias was found to serve as the core cognitive mechanism of depression disorder. However, there was no evidence to show the reason lead to negative bias. In the current study, investigators hypothesized that the blurring self representation was the neural correlates in depression disorder.

DETAILED DESCRIPTION:
To test investigators' hypothesis, investigators adopted the self-referential task and fMRI to investigate the neural representation of self in depression patients, and compared with healthy control.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be clinical diagnosis of major depression disorder.
* Healthy control participants should be age-matched with depression group, and should have no history of neurological or psychiatric diagnoses

Exclusion Criteria:

* Patients who also have bipolar disorder, schizophrenia, anxiety disorder
* Healthy controls who have history of mental disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with depression and healthy control
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Neural representation of self | through study completion, an average of 2 year
  We adopted the self referential task. In the task, participants were asked to judge whether a given word was appropriate to describe oneself (self-judgement condition), a celebrity (other-judgement condition) by pressing one of the two buttons with the index or middle finger. For judgments of each target person (i.e, self and celebrity), there were 3 categories of words describing the mental (personality traits, such as hard-working, friendly), physical (physical attributes, such as black hair, big eyes) and social (social roles, such as student, American) dimension of person knowledge. The fMRI task contained 6 runs, with 4.6 minutes per run.
  This paradigm and task allowed us to investigated the neural representation of self by comparing the BOLD activity under self-judgement condition with BOLD activity under other-judgement condition.

IPD SHARING:
Plan to Share IPD: No